CLINICAL TRIAL: NCT02215941
Title: A Randomized, Double Blind, Placebo-Controlled, Parallel Group, Dose Escalation Study to Characterize the Pharmacokinetics and Safety of 8% TV-45070 Ointment Following 7.5 Days of Twice Daily Topical Application in Healthy Subjects
Brief Title: Study to Characterize the Pharmacokinetics and Safety of TV-45070 Ointment in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: TV45070-PK-10033
Record Dates: First submitted 2014-08-06; First posted 2014-08-13 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — TV-45070

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- TV-45070 7% (Experimental): twice daily topical application to 7% body surface area for 7.5 days (15 applications)
  Interventions: Drug: TV-45070
- TV-45070 21% (Experimental): twice daily topical application to 21% body surface area for 7.5 days (15 applications)
  Interventions: Drug: TV-45070
- TV-45070 53% (Experimental): twice daily topical application to 53% body surface area for 7.5 days (15 applications)
  Interventions: Drug: TV-45070
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TV-45070 — TV-45070 8% ointment
  Arms: TV-45070 21%; TV-45070 53%; TV-45070 7%
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to characterize the pharmacokinetics of TV-45070 in plasma following single and multiple-dose topical application of 8% TV-45070 ointment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects aged 18 to 50 years
* Body Mass Index (BMI) ≥18.0 and ≤32.0 kg/m2.
* Able and willing to provide written informed consent.
* Able and willing to comply with all study procedures and restrictions.

Exclusion Criteria:

* History or evidence of clinically significant illness or surgery
* Presence of open wounds, sunburn, tattoo, major scarring, non-intact or damaged in the proposed application area that would interfere with the application of the study drug treatments or biopsies.
* History of significant drug or alcohol abuse
* Use of prescription drugs within 30 days or 5 half-lives (whichever is longer) prior to Day 1.
* Use of topical application of an OTC medicated or prescription medication or other skin creams/ointments (eg, moisturizers, balms) in the areas intended for study drug administration within 7 days prior to Day 1. Use of topical capsaicin within 6 months prior to Day 1.
* Pregnant or nursing females
* Shaving or waxing the planned study treatment application area within 7 days prior Day 1.
* Laser hair removal of the planned study treatment application area within 2 months prior to Day 1.

  * other criteria apply, please contact the investigator for more information

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations | Day 8

SECONDARY OUTCOMES:
Drug level in skin | Days 1, 8, 15, 22, 29
Excretion of drug in urine | Day 8
Identification of metabolites in blood | Days 8, 10
Identification of metabolites in urine | Day 8
Identification of metabolites in skin | Days 1, 8, 15, 22, 29
Intraepidermal nerve fiber density in skin | Days 1, 8, 15, 29
Percentage of Participants with Adverse Events | 10 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (1):
- Teva Investigational Site 12961, Lenexa, Kansas, United States